CLINICAL TRIAL: NCT01462175
Title: A Multi-center, Open Label, First in Human Phase I Dose Escalation Study of Single Agent RO5503781, a Small Molecule MDM2 Antagonist, Administered Orally in Patients With Advanced Malignancies, Except Leukemia
Brief Title: A First-In-Human Study of RO5503781 in Participants With Advanced Malignancies Except Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP27872; 2011-002767-15 (EudraCT Number)
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Schedule A: RO5503781 QW (Experimental): Participants will receive multiple ascending doses of RO5503781 orally once weekly (QW) x 3 followed by 13 days of rest in a 28 days cycle.
  Interventions: Drug: RO5503781
- Schedule B: RO5503781 QD (Experimental): Participants will receive multiple ascending doses of RO5503781 orally QD x 5 followed by 13 days of rest in a 28 days cycle.
  Interventions: Drug: RO5503781

INTERVENTIONS:
Drug: RO5503781

SUMMARY:
This multicenter, open label, dose-escalating study will evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of RO5503781, administered once daily (QD) or once weekly (QW) in participants with advanced malignancies except leukemia. Participants will receive multiple escalating oral doses in two different dosing schedules (Sch) until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced malignancies, except all forms of leukemia, for which standard curative or palliative measures do not exist, are no longer effective, or are not acceptable to the participants
* Measurable disease (according to RECIST or Cheson criteria) or evaluable disease prior to administration of study drug
* Minimum weight of 35 kg and life expectancy of greater than or equal to (>=) 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Acute toxicities from any prior anti-tumor therapy, surgery, or radiotherapy must have resolved to NCT-CTCAE Grade less than or equal to (<=) 1
* Adequate renal, hepatic and bone marrow function
* Participants with stable Central Nervous System (CNS) metastasis and with chronic, stable and rate controlled atrial fibrillation
* Participants in consideration for the biomarker cohorts or apoptosis imaging cohort must consent and be able to undergo paired biopsies for tumor biomarker analyses
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* History of any form of leukemia except for Stage 0 and 1 chronic lymphocytic leukemia (CLL) not requiring treatment in addition to the underlying solid tumor
* Use of hormonal therapy within 2 weeks and use of other investigational agents or having received investigational drugs <= 4 weeks prior to study treatment start
* History of seizure disorders or unstable CNS metastases
* Severe and/or uncontrolled cardiovascular disease or disorder
* Active (acute or chronic) or uncontrolled infection
* Pregnant or breastfeeding women
* HIV-positive participants who are currently receiving anti-retroviral treatment
* Known coagulopathy, platelet disorder or history of non-drug induced thrombocytopenia
* Participants receiving oral or parenteral anticoagulants/antiplatelet agents; anticoagulant flushes for maintenance of indwelling catheters are allowed
* Participants with known bone marrow disorder which may interfere with bone marrow recovery
* Participants with hypersensitivity reaction to 18Fluorothymidine (FLT or 18F) compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 28 days
Percentage of Participants With Dose Limiting Toxicities (DLTs) | up to 28 days
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | approximately 1.5 years

SECONDARY OUTCOMES:
Plasma Concentration of RO5503781 | Sch A: pre-dose (PrD; 0 hour), 1, 2, 3, 4, 6, 8, 12 hours post-dose (PoD) on Day 1, 15; PrD (0 hour) on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Urine Concentration of RO5503781 | Schedule A and B: Pre-dose, 0-4, 4-8, 8-12, 12-24 hours post-dose on Day 1, Day 2
Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Percentage of Participants With Objective Response [Complete Response (CR) plus Partial Response(PR)] According to Response Evaluation Criteria in Solid Tumors (RECIST) | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Standardized Uptake Value (SUV) obtained from the Positron Emission Tomography With 18-Fluorothymidine [(18F)-FLT-PET) Images | Baseline, Cycle1 Day 5, Cycle 3 Day 1
Pharmacodynamics: p21 Levels in Tumor as Measured by Immunohistochemistry | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Tumor suppressor gene (p53) Levels in Tumor as Measured by Immunohistochemistry | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Murine Double Minute 2 (MDM2) Levels in Tumor as Mesured by Reverse transcription polymerase chain reaction (RT-PCR) | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Ki-67 Levels in Tumor as Measured by Immunohistochemistry | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL) Levels in Tumor as Measured by Immunohistochemistry | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Progression Free Survival (PFS) According to Cheson Criteria | andomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: p53 Mutation Status in Tumor as Measured by AmpliChip p53 Test | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Mouse Double Minute 2 Homolog (MDM2) Gene Copy Number in Tumor as Measured by in situ Hybridization | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | PrD (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours PoD on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Area Under the Curve From Time Zero to Extrapolated 168 hours [AUC(0-168)] | Prd (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Maximum Observed Plasma Concentration (Cmax) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Maximum Observed Plasma Concentration (Cmax) | PrD (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Time to Reach Maximum Observed Plasma Concentration (Tmax) | PrD (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Plasma Decay Half-Life (t1/2) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Plasma Decay Half-Life (t1/2) | PrD (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Terminal Elimination Rate Constant (Kel) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Food-Effect: Terminal Elimination Rate Constant (Kel) | PrD (0 hour), 1, 2, 3, 4, 6, 8 and 12 hours post-dose on Day 1, 8, 15; on Day 2, 3, 4/5, 6/7, 9, 10, 11/12, 13/14, 16, 17, 18/19, 20/21, 22
Apparent Oral Clearance (CL/F) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Apparent Volume of Distribution (Vz/F) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12
Percentage of Participants With Objective Response [Complete Response (CR) plus Partial Response(PR)] According to Cheson Criteria | Randomization until progressive disease or death (assessed at baseline and every 8 weeks thereafter until progressive disease, death or end of study [up to approximately 1.5 years])
Pharmacodynamics: Macrophage Inhibitory Cytokine 1 (MIC-1) Levels in Blood as Measured by Enzyme-linked Immunosorbent Assay (ELISA) | Sch A: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 15; PrD on Day 8; on Day 2, 3, 4/5, 6/7, 16, 17, 18/19, 20/21, 22; Sch B: PrD (0 hour), 1, 2, 3, 4, 6, 8, 12 hours PoD on Day 1, 5; Day 6, 7, 8/9, 10/11, 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Melbourne, Victoria, Australia
- Canada (3):
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (2):
  - Bordeaux
  - Lyon
- Groningen, Netherlands
- Seoul, South Korea

REFERENCES:
- [Derived] Italiano A, Miller WH Jr, Blay JY, Gietema JA, Bang YJ, Mileshkin LR, Hirte HW, Higgins B, Blotner S, Nichols GL, Chen LC, Petry C, Yang QJ, Schmitt C, Jamois C, Siu LL. Phase I study of daily and weekly regimens of the orally administered MDM2 antagonist idasanutlin in patients with advanced tumors. Invest New Drugs. 2021 Dec;39(6):1587-1597. doi: 10.1007/s10637-021-01141-2. Epub 2021 Jun 28. PMID 34180037